CLINICAL TRIAL: NCT05992584
Title: Lenvatinib, Sintilimab Plus Y-90 Selective Internal Radiation Therapy for Patients With Unresectable Intermediate-advanced Hepatocellular Carcinoma: a Prospective, Single-center, Single Arm Trial
Brief Title: Lenvatinib, Sintilimab Plus SIRT for Unresectable HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIIR-14
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Lenvatinib; Sintilimab; Yttrium-90
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; sintilimab; Sirtuins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Len-Sin-SIRT (Experimental): Lenvatinib, sintilimab plus SIRT
  Interventions: Drug: Lenvatinib, sintilimab plus SIRT

INTERVENTIONS:
Drug: Lenvatinib, sintilimab plus SIRT — Lenvatinib 12mg (body weight ≥60kg) or 8mg (body weight <60kg) P.O. QD and sintilimab 200mg I.V. q3w will be started at 3-7 days after the first SIRT. Treatment of sintilimab will last up to 24 months. Patients will be allowed to have lenvatilib or sintilimab as a sigle agent and will be still considered on study when the other drug cause intolerable toxicity.

SUMMARY:
This study is conducted to evaluate the efficacy and safety of lenvatinib, sintilimab plus Y-90 selective internal radiation therapy (SIRT) for patients with unresectable intermediate-advanced hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
This is a single-center, prospective study to evaluate the efficacy and safety of lenvatinib, sintilimab plus SIRT (Len-Sin-SIRT) in patient with unresectable HCC.

30 patients with unresectable intermediate-advanced HCC (BCLC B/C stage) will be enrolled in this study. The patients will receive lenvatinib (body weight ≥60kg, 12mg; body weight <60kg, 8mg; P.O. QD) and sintilimab (200mg I.V. Q3W) at 3-7 days after SIRT. Sintilimab will last up to 24 months, or until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. Lenvatinib will last until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first.

The primary end point of this study is Progression free survival (PFS) per mRECIST. The secondary endpoints are PFS per RECIST 1.1, objective response rate (ORR), disease control rate (DCR), overall survival (OS) and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Unresectable HCC (BCLC stage B/C) with diagnosis confirmed by histology/cytology or clinically
* At least one measurable untreated lesion
* Intrahepatic tumors can be treated with 1-2 session of SIRT
* Child-Pugh score 5-7
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1
* Life expectancy of at least 3 months
* Patients with active hepatitis B are allowed, but they need to receive antiviral treatment to achieve a HBV DNA<10^3 IU/mL
* Patients with hepatitis C need to finish the anti-HCV treatment

Exclusion Criteria:

* tumor extent ≥70% liver occupation
* Tumor thrombus involving main portal vein or both the first left and right branch of portal vein
* Vena cava invasion
* Central nervous system metastasis
* Metastatic disease that involves major airways or blood vessels
* Patients who previously received hepatic arterial infusion chemotherapy (HAIC), transarterial chemoembolization (TACE), transarterial embolization (TAE), radiotherapy, systemic therapy, or immunotherapy for HCC
* History of organ and cell transplantation
* Prior esophageal and/or gastric varices bleeding
* History of hepatic encephalopathy
* Peripheral blood white blood cell count<3×10^9/L, platelet count<50×10^9/L
* Prolongation of prothrombin time ≥ 4 seconds
* Severe organ dysfunction (heart, lungs, kidneys)
* History of malignancy other than HCC
* HBsAg and anti-HCV antibody positive concurrently
* Human immunodeficiency virus (HIV) infected

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2026-01-09 (Estimated); Study Completion 2026-08-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) according to mRECIST | 2.5 years
  The time from initiation of treatment until the first occurrence of disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression free survival (PFS) according to RECIST 1.1 | 2.5 years
  The time from initiation of treatment until the first occurrence of disease progression or death from any cause, whichever occurs first.
Objective response rate (ORR) | 2.5 years
  The percentage of patients who had a best overall tumor response rating of complete response (CR) or partial response (PR) according to mRECIST and RECIST 1.1
Disease control rate (DCR) | 2.5 years
  The percentage of patients who had a tumor response rating of CR, PR, or stable disease (SD) according to mRECIST and RECIST 1.1
Overall survival (OS) | 2.5 years
  The time from initiation of treatment until the date of death from any cause.
Adverse Events (AEs) | 2.5 years
  Number of patients with AEs assessed by NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided